CLINICAL TRIAL: NCT04682158
Title: Propranolol With Standard Chemoradiation for Esophageal Adenocarcinoma A Phase II Study
Brief Title: Propranolol With Standard Chemoradiation for Esophageal Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: I 630420
Record Dates: First submitted 2020-12-21; First posted 2020-12-23 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Esophageal Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — Carboplatin; Radiotherapy, Conformal; Radiation; Propranolol; propranolol CR; Radiotherapy, Intensity-Modulated; Paclitaxel; Taxes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Chemoradiation Therapy - Group I (Active Comparator): Patients receiving beta-blockers undergo radiation therapy in the form of IMRT or 3D CRT over 23-28 fractions for 5 days per week (Monday-Friday) for 5 weeks, and receive paclitaxel IV QW and carboplatin IV QW for 5 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Radiation: 3 Dimensional Conformal Radiation Therapy; Radiation: Intensity Modulated Radiation Therapy; Drug: Paclitaxel
- Chemoradiation Therapy - Group II (Active Comparator): Patients undergo CRT as in Group I in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: 3 Dimensional Conformal Radiation Therapy
- Chemoradiation Therapy plus Propanolol (Experimental): Patients undergo radiation therapy as in Group I. Patients receive propranolol PO BID for 4-8 weeks while receiving standard neoadjuvant/definitive chemotherapy or chemotherapy-immunotherapy or CRT in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: 3 Dimensional Conformal Radiation Therapy; Drug: Propranolol; Radiation: Intensity Modulated Radiation Therapy

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: (SP-4-2)-diammine[1,1-cyclobutanedicarboxylato(2--)-O,O'']platinum; Blastocarb; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Ribocarbo
  Arms: Chemoradiation Therapy - Group I
Radiation: 3 Dimensional Conformal Radiation Therapy — Undergo 3D CRT
  Other Names: 3D-CRT; Radiation
Drug: Propranolol — Subject will be treated with 30 mg po BID Propranolol for up to 6 weeks
  Other Names: 2-Propanol-1-[(1-methylethyl)amino]-3-(1-naphthalenyloxy) Hydrochloride; 318-98-9; Inderal; Innopran XL
  Arms: Chemoradiation Therapy plus Propanolol
Radiation: Intensity Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT
  Arms: Chemoradiation Therapy - Group I; Chemoradiation Therapy plus Propanolol
Drug: Paclitaxel — Given IV
  Other Names: 33069-62-4; 5Beta,20-epoxy-1,2alpha; Anzatax; Bristaxol; Praxel; Taxol
  Arms: Chemoradiation Therapy - Group I

SUMMARY:
This phase II trial studies the side effects and best dose of propranolol when administered concurrently with SOC neoadjuvant CRT in patients with esophageal carcinoma, with a safety lead-in and dose expansion cohort. Patients who are already on β-blockers will receive standard of care CRT, or definitive chemotherapy or chemotherapy-immunotherapy and will be considered separately as a single arm prospective cohort

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and efficacy of propranolol hydrochloride (propranolol) in combination with standard neoadjuvant/definitive chemotherapy or chemotherapy-immunotherapy or chemoradiation therapy (CRT) for esophageal cancer.

SECONDARY OBJECTIVE:

I. To estimate overall survival (OS) and pathologic response rate in patients that undergo surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing definitive or neoadjuvant CRT for histologically confirmed esophageal adenocarcinoma
* Have an ECOG performance status of 0-1
* Have the ability to swallow and retain oral medication. If a patient is not able to swallow, they are still eligible for study provided they have an enteric feeding placed which will permit administration of crushed tablets or liquid formula propranolol prior to first radiation treatment
* Participants of child-bearing potential must have a negative pregnancy test at study entry And then agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. - Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* Contraindications to the use of beta-blockers, e.g.; uncontrolled depression, unstable angina pectoris, uncontrolled heart failure (New York Heart Association (NYHA) Grade III or IV), hypotension ( systolic blood pressure <100 mmHg), severe asthma or COPD, uncontrolled type I or type II diabetes mellitus (HbA1C >8.5 or fasting plasma glucose > 160 mg/dL at screening), symptomatic peripheral arterial disease or Raynaud's syndrome, untreated pheochromocytoma, current calcium channel blocker use (Non-dihydropyridines such as verapamil) or rhythm control agents such as digoxin and amiodarone. Patients with pacemakers will be excluded
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection,symptomatic congestive heart failure, unstable angina pectoris, psychiatric illness/social situations that would limit compliance with study requirements, cardiac arrhythmia (atrial fibrillation/flutter), severe bradycardia (heart rate of <50 beats per minute or 1st/ 2nd /3rd degree heart block)
* Pregnant or nursing female participants,
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Adverse Events | Up to 5 years
  To determine the safety and efficacy of the combination of propranolol plus chemoradiation
Progression Free Survival | UP to 5 years
  Imaging findings from first radiation treatment to progression of disease

SECONDARY OUTCOMES:
Overall Survival | Up to 5 years
  will be assessed by chart review of date of last follow-up or date of death

CONTACTS AND LOCATIONS:
Overall Officials: Anurag Singh, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided